CLINICAL TRIAL: NCT04800289
Title: Evaluation of Patient Satisfaction and Therapeutic Impact Regarding Joint Consultation Rheumatologist/Dermatologist
Acronym: RHUMPSO
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Other Study IDs: CHM-2019/S7/11
Record Dates: First submitted 2021-03-12; First posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaires — questionnaires about disease and satisfaction of patient

SUMMARY:
Current increase in the number of multidisciplinary consultations, but little documentation on their impact on patient management. More specifically, in the context of psoriatic arthritis, we are seeking to investigate the interest for the patient, through his or her satisfaction and the evolution of the activity of his or her pathology, of a global, joint management in Rheumatology and Dermatology.

ELIGIBILITY:
Inclusion Criteria:

* All patients received in a joint rheumatologist/dermatologist consultation at the Le Mans Hospital

Exclusion Criteria:

* Diagnosis of psoriatic arthritis not retained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients received in a joint rheumatologist/dermatologist consultation at the Le Mans Hospital
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-07-19 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
impact on patient satisfaction and the evolution of their pathology of these mixed consultations, Dermatologist and Rheumatologist, in the context of psoriatic arthritis. | 5 years after inclusion
  evaluate the impact on patient satisfaction and the evolution of their pathology of these mixed consultations, Dermatologist and Rheumatologist, in the context of psoriatic arthritis.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Du Mans, Le Mans, France

IPD SHARING:
Plan to Share IPD: No